CLINICAL TRIAL: NCT06189274
Title: Anatomy-Based Cochlear Implant Array Selection for Patients With Single-Sided Deafness
Brief Title: Anatomy Based Selection of CI Array for SSD Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nova Scotia Health Authority (Other)
Collaborators: Med-El Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NSHSCMEDEL
Record Dates: First submitted 2023-12-18; First posted 2024-01-03 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Single-Sided Deafness

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Anatomy-Based Electrode Selection (Experimental): For individuals in the anatomy-based electrode (ABE) group, magnetic resolution imaging (MRI) or computed tomography (CT) scans will be evaluated by MED-EL Canada employees. Based on these results, an appropriate electrode array will be selected.
  Interventions: Other: Anatomy-Based Electrode Array Selection
- Standard of Care Electrode Selection (Active Comparator): The comparison in this study will be to current standard of care, which is to select a single electrode length for most patients, in this case the FLEX28 electrode, which is 28 mm long.
  Interventions: Other: Standard of Care Electrode Array Selection

INTERVENTIONS:
Other: Anatomy-Based Electrode Array Selection — Use of pre-operative imaging to select the appropriate length electrode vs standard of care
  Other Names: OTOPLAN
  Arms: Anatomy-Based Electrode Selection
Other: Standard of Care Electrode Array Selection — Use of standard of care electrode which is the FLEX 28 electrode
  Arms: Standard of Care Electrode Selection

SUMMARY:
The purpose of the study is to evaluate cochlear implant speech outcomes and subjective benefit for cochlear implant recipients with single-sided deafness using patient-specific, anatomy-based array selection versus standard of care with a fixed array size for all patients. Subjects will prospectively be assigned to receive an Anatomy-Based Electrode (FLEX26, FLEX28, or FLEXSOFT) or the Standard of Care Electrode array (FLEX28). Speech performance and subjective benefit will be evaluated between these two groups.

DETAILED DESCRIPTION:
To determine the effectiveness of Anatomy-Based Electrode selection versus Standard of Care Electrode selection in SSD listeners a prospective, single-blinded study design will be used to evaluate the outcomes in these two groups by evaluating speech understanding in quiet, speech understanding in noise, subjective listening difficulty and sound quality, and datalogging.

Subjects will be randomly assigned to either group to receive an electrode based on their anatomy (ABE) or the Standard of Care electrode (SOCE). Five participants will be in each group, for a total of 10 participants.

All subjects will receive a MED-EL Cochlear Implant and will subsequently be fit with an audio processor approved by Health Canada. Post-operative evaluations will occur at one and six months post-activation.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older at the time of implantation
* Unilateral severe to profound sensorineural hearing loss, as defined by a pure-tone average (500, 1000, 2000, and 4000 Hz) of 70 dB HL or greater
* Normal hearing mild hearing loss in the non-implanted ear, as defined by a pure-tone average (500, 1000, 2000, and 4000 Hz) of 40 dB or less
* Deemed an appropriate candidate by the investigator
* Fluent in English

Exclusion Criteria:

* Duration of profound hearing loss of 10 years or more
* Sudden onset of hearing loss within six months of implantation
* Evidence of non-functional cochlear nerve using appropriate imaging modality to be determined by the investigator
* Other retrocochlear hearing loss
* Evidence of severe cochlear malformation (i.e., common cavity or ossification)
* External or middle ear infection
* Suspected developmental or cognitive concern
* Other medical contraindication for surgery or anesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Speech perception in spatially separated noise | 6 months post activation
  Change in percent correct on the AzBio sentences in noise, with speech presented to the front and noise to the better hearing ear

SECONDARY OUTCOMES:
Speech perception in noise | 6 months post activation
  Change in percent correct on the AzBio sentences in noise, in two conditions. Condition 1 is with speech and noise both presented to the front. Condition 2 is with speech presented from the front and noise presented to the CI ear
Speech perception in quiet | 6 months post activation
  Change in percent correct on the CNC words in quiet in implanted ear.
Speech Spatial and Qualities of Hearing Scale (SSQ) | 6 months post activation
  Subjective questionnaire on speech perception and sound quality
Datalogging | 6 months post activation
  Evaluate average daily device use

IPD SHARING:
Plan to Share IPD: No